CLINICAL TRIAL: NCT02814175
Title: A Phase 4 Open-label Randomized Controlled Study COmparing the Effectiveness of Adalimumab iNTROduction and Methotrexate Dose escaLation in Subjects With Psoriatic Arthritis (CONTROL)
Brief Title: A Study of Subjects With Psoriatic Arthritis to Investigate the Effectiveness of Adalimumab Introduction Compared With Methotrexate Dose Escalation (CONTROL)
Acronym: CONTROL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M14-496; 2016-000191-21 (EudraCT Number)
Record Dates: First submitted 2016-06-21; First posted 2016-06-27 (Estimated); Results first posted 2020-11-23 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-10

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Methotrexate; Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Part 1: MTX Escalated Dose (Active Comparator): Methotrexate (MTX) escalated to 20 - 25 mg or highest tolerable dose every week (ew)
  Interventions: Drug: methotrexate (MTX)
- Part 1: ADA + MTX (Experimental): Adalimumab (ADA) 40 mg every other week (eow) in combination with MTX 15 mg ew
  Interventions: Drug: methotrexate (MTX); Biological: adalimumab (ADA)
- Part 2: MTX Escalated Dose (Active Comparator): Participants achieving minimal disease activity (MDA) at Week 16 on MTX escalated to 20 -25 mg or highest tolerable dose ew, continued with the same MTX dose
  Interventions: Drug: methotrexate (MTX)
- Part 2: ADA + MTX Escalated Dose (Active Comparator): Participants not achieving MDA at Week 16 on MTX escalated to 20 - 25 mg or highest tolerable dose ew, received ADA 40 mg eow in combination with MTX 20 - 25 mg or highest tolerable dose ew
  Interventions: Drug: methotrexate (MTX); Biological: adalimumab (ADA)
- Part 2: ADA (Experimental): Participants achieving MDA at Week 16 on ADA 40 mg eow plus MTX 15 mg ew, had MTX completely withdrawn at Week 16 and continued receiving ADA as monotherapy
  Interventions: Biological: adalimumab (ADA)
- Part 2: ADA ew + MTX (Experimental): Participants not achieving MDA at Week 16 on ADA 40 mg eow plus MTX 15 mg ew, had ADA escalated to 40 mg ew in combination with MTX 15 mg ew
  Interventions: Drug: methotrexate (MTX); Biological: adalimumab (ADA)

INTERVENTIONS:
Drug: methotrexate (MTX)
  Arms: Part 1: ADA + MTX; Part 1: MTX Escalated Dose; Part 2: ADA + MTX Escalated Dose; Part 2: ADA ew + MTX; Part 2: MTX Escalated Dose
Biological: adalimumab (ADA)
  Arms: Part 1: ADA + MTX; Part 2: ADA; Part 2: ADA + MTX Escalated Dose; Part 2: ADA ew + MTX

SUMMARY:
An interventional Phase 4 open-label, randomized, controlled, parallel-group, multi-country study in participants with psoriatic arthritis (PsA) consisting of 2 parts: Part 1 (Day 1 up to Week 16) is designed to compare the achievement of minimal disease activity (MDA) between participants randomized to either adalimumab in combination with methotrexate (MTX) or MTX alone escalated to the highest recommended or tolerable dose; Part 2 (Week 16 through Week 32) is designed to evaluate the maintenance or achievement of MDA on 4 different treatment regimens using adalimumab and/or MTX, with participant allocation based on the initial randomized treatment and achievement of MDA in Part 1, and with rescue treatment option.

ELIGIBILITY:
Inclusion Criteria:

1. PsA diagnosis established at least 4 weeks prior to the date of the Screening visit and confirmed by ClASsification of Psoriatic Arthritis (CASPAR) criteria
2. Not in MDA at the time of screening
3. Has 3 or more tender and 3 or more swollen joints
4. Treated with methotrexate 15 mg (weekly) for at least 4 weeks

Exclusion Criteria:

1. Contraindications to adalimumab therapy and/or known hypersensitivity to adalimumab or its excipients
2. History of methotrexate intolerance/toxicity
3. Medical conditions(s) precluding methotrexate dose increase above 15 mg
4. Had prior exposure to any tumor necrosis factor (TNF) inhibitor, other mechanism of action biologic DMARD (bDMARD) or any systemic biologic agent in general

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2016-08-05 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2020-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (60):
- United States (12):
  - AZ Arthritis & Rheum Research /ID# 161796, Sun City, Arizona
  - LeJenue Research Associates /ID# 200093, Miami, Florida
  - Deerbrook Medical Associates /ID# 158655, Vernon Hills, Illinois
  - Ochsner Clinic Foundation /ID# 155178, Baton Rouge, Louisiana
  - Clinical Pharmacology Study Gr /ID# 161057, Worcester, Massachusetts
  - Shores Rheumatology, PC /ID# 162697, Saint Clair Shores, Michigan
  - Coastal Carolina Health Care /ID# 152088, New Bern, North Carolina
  - PMG Research of Wilmington LLC /ID# 152089, Wilmington, North Carolina
  - Altoona Ctr Clinical Res /ID# 152087, Duncansville, Pennsylvania
  - Metroplex Clinical Research /ID# 162486, Dallas, Texas
  - Swedish Medical Center /ID# 162051, Seattle, Washington
  - West Virginia Research Inst /ID# 157815, South Charleston, West Virginia
- Australia (5):
  - Royal Prince Alfred Hospital /ID# 153144, Camperdown, New South Wales
  - Optimus Clinical Research Pty. /ID# 153145, Kogarah, New South Wales
  - Liverpool Hospital /ID# 153147, Liverpool, New South Wales
  - BJC Health /ID# 153875, Paramatta, New South Wales
  - Box Hill Hospital /ID# 153146, Melbourne, Victoria
- Brazil (2):
  - Hospital de Clinicas de Porto Alegre /ID# 152345, Porto Alegre, Rio Grande do Sul
  - Faculdade de Medicina do ABC /ID# 152344, Santo André, São Paulo
- Bulgaria (2):
  - MHAT Trimontsium /ID# 152658, Plovdiv
  - Diag Consult Ctr 17 Sofia EOOD /ID# 152657, Sofia
- Canada (8):
  - Rheumatology Research Assoc /ID# 161600, Edmonton, Alberta
  - Percuro Clinical Research, Ltd /ID# 161601, Victoria, British Columbia
  - Manitoba Clinic /ID# 151939, Winnipeg, Manitoba
  - St. Clare's Mercy Hospital /ID# 159680, St. John's, Newfoundland and Labrador
  - The Waterside Clinic /ID# 151938, Barrie, Ontario
  - Adachi Medicine Prof. Corp /ID# 152575, Hamilton, Ontario
  - Ctr. de Rheum de l'est du QC /ID# 151937, Rimouski, Quebec
  - Groupe de Recherche en Maladies Osseuses /ID# 205693, Sainte-Foy, Quebec
- Colombia (3):
  - Centro de Investigacion en Reumatologia y Especialidades Medicas- CIREEM SAS /ID# 151954, Bogota, Cundinamarca
  - Riesgo de Fractura S.A - CAYRE /ID# 153817, Bogotá
  - San Vicente Fundacion /Id# 171324, Medellín
- Czechia (2):
  - Revmatolog s.r.o. /ID# 151753, Jihlava, Jihlava
  - Nuselská poliklinika, Revmatologie /ID# 151754, Prague, Praha 4
- Germany (5):
  - Universitaetsklinik Heidelberg /ID# 152229, Heidelberg, Baden-Wurttemberg
  - Fachpraxis fuer Rheumatologie und Osteologie /ID# 203982, Bruchhausen-Vilsen, Lower Saxony
  - Univ Hosp Schleswig-Holstein, Campus Kiel, Klinik furer Innere Medizin /ID# 152231, Kiel, Schleswig-Holstein
  - CIRI GmbH /ID# 152228, Frankfurt
  - Hamburger Rheuma I /ID# 164055, Hamburg
- Italy (3):
  - Universita di Catanzaro Magna Graecia /ID# 152013, Catanzaro, Calabria
  - Azienda Ospedaliera Policlinic /ID# 152011, Rome
  - A.O. Universitaria Senese /ID# 152012, Siena
- Poland (4):
  - McBk Sc /Id# 163089, Grodzisk Mazowiecki, Masovian Voivodeship
  - Centrum Medyczne AMED /ID# 164047, Warsaw, Masovian Voivodeship
  - SANUS Szpital Specjalistyczny /ID# 151988, Stalowa Wola, Podkarpackie Voivodeship
  - ClinicMed Badurski i wspolnicy SJ /ID# 151987, Bialystok
- Puerto Rico (2):
  - Dr. Ramon L. Ortega-Colon, MD /ID# 152957, Carolina
  - GCM Medical Group, PSC /ID# 152091, San Juan
- Hamad Hospital /ID# 152334, Doha, Baladīyat ad Dawḩah, Qatar
- Spain (6):
  - Corporac Sanitaria Parc Tauli /ID# 151759, Sabadell, Barcelona
  - Hospital Univ Germans Trias I Pujol /ID# 151760, Badalona
  - Hospital Universitario Reina S /ID# 151761, Córdoba
  - Hospital Manises /ID# 162778, Manises
  - Hospital Univ Canarias /ID# 206489, Santa Cruz de Tenerife
  - Hospital de Viladecans /ID# 163875, Viladecans
- United Kingdom (5):
  - Royal National Hosp for Rheuma /ID# 152767, Bath
  - Western General Hospital /ID# 155195, Edinburgh
  - Altnagelvin Area Hospital /ID# 152766, Londonderry
  - Central Manchester University /ID# 152765, Manchester
  - Lancashire Care NHS Foundation /ID# 152769, Preston

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Coates LC, Tillett W, D'Agostino MA, Rahman P, Behrens F, McDearmon-Blondell EL, Bu X, Chen L, Kapoor M, Conaghan PG, Mease P. Comparison between adalimumab introduction and methotrexate dose escalation in patients with inadequately controlled psoriatic arthritis (CONTROL): a randomised, open-label, two-part, phase 4 study. Lancet Rheumatol. 2022 Apr;4(4):e262-e273. doi: 10.1016/S2665-9913(22)00008-X. Epub 2022 Feb 25. PMID 38288922

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 246 participants randomized; 1 participant did not receive study medication. Upon completion of Part 1, eligible participants continued to Part 2, so no additional participants were enrolled in Part 2.
Pre-assignment Details: Intent-To-Treat Part 1 (ITT Part 1) population comprised all participants randomized and received at least 1 dose of study medication in Part 1. ITT Long Term (ITT LT) population included all participants who continued to Part 2 and received at least 1 dose of Part 2 study medication; no additional participants were enrolled into Part 2.
Groups:
- Part 1: ADA + MTX: Adalimumab (ADA) 40 mg every other week (eow) in combination with methotrexate (MTX) 15 mg every week (ew)
- Part 2: MTX Escalated Dose: Participants achieving minimal disease activity (MDA) at Week 16 on methotrexate (MTX) escalated to 20 -25 mg or highest tolerable dose every week (ew), continued with the same MTX dose
- Part 2: ADA +MTX Escalated Dose: Participants not achieving minimal disease activity (MDA) at Week 16 on methotrexate (MTX) escalated to 20 - 25 mg or highest tolerable dose every week (ew), received adalimumab (ADA) 40 mg every other week (eow) in combination with MTX 20 - 25 mg or highest tolerable dose ew
- Part 2: ADA: Participants achieving minimal disease activity (MDA) at Week 16 on adalimumab (ADA) 40 mg every other week (eow) plus methotrexate (MTX) 15 mg every week (ew), had MTX completely withdrawn at Week 16 and continued receiving ADA as monotherapy
- Part 2: ADA ew + MTX: Participants not achieving minimal disease activity (MDA) at Week 16 on adalimumab (ADA) 40 mg every other week (eow) plus methotrexate (MTX) 15 mg every week (ew), had ADA escalated to 40 mg ew in combination with MTX 15 mg ew
Period: Part 1
Arm/Group | Part 1: MTX Escalated Dose | Part 1: ADA + MTX | Part 2: MTX Escalated Dose | Part 2: ADA +MTX Escalated Dose | Part 2: ADA | Part 2: ADA ew + MTX
Started | 122 | 123 | 0 | 0 | 0 | 0
Completed | 110 | 117 | 0 | 0 | 0 | 0
Not Completed | 12 | 6 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 3 | 0 | 0 | 0 | 0
Not completed — Withdrawal Consent | 8 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 2 | 0 | 0 | 0 | 0
Period: Part 2
Arm/Group | Part 1: MTX Escalated Dose | Part 1: ADA + MTX | Part 2: MTX Escalated Dose | Part 2: ADA +MTX Escalated Dose | Part 2: ADA | Part 2: ADA ew + MTX
Started | 0 | 0 | 15 | 95 | 54 | 63
Completed | 0 | 0 | 15 | 91 | 52 | 57
Not Completed | 0 | 0 | 0 | 4 | 2 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1 | 2
Not completed — Withdrawal Consent | 0 | 0 | 0 | 2 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: The Intent-To-Treat Part 1 (ITT Part 1) population comprises all participants who were randomized and received at least one dose of the study medication during Part 1.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: MTX Escalated Dose | Part 1: ADA + MTX | Total
Number analyzed (Participants) | 122 | 123 | 245
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (12.69) | 51.4 (12.23) | 50.1 (12.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 64 | 123
  Male | 63 | 59 | 122
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 27 | 54
  Not Hispanic or Latino | 95 | 96 | 191
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 1 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 2 | 2 | 4
  White | 111 | 115 | 226
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Minimal Disease Activity (MDA) (Non-responder Imputation [NRI]) (Part 1)
Description: Minimal disease activity (MDA) for psoriatic arthritis (PsA) was defined as fulfilling at least 5 of the following 7 criteria: tender and swollen joint counts (TJC) ≤ 1 (out of TJC68 assessed in this study), swollen joint count (SJC) ≤ 1 (out of SJC66 assessed in this study), Psoriasis Area and Severity Index (PASI) ≤ 1 or body surface area (BSA) ≤ 3; Patient's assessment of pain visual analogue scale (VAS) ≤ 15, Patient's global assessment of disease activity (PtGA) VAS ≤ 20, Health Assessment Questionnaire Disability Index (HAQ-DI) score ≤ 0.5, and tender entheseal points ≤ 1 (out of 8 assessed in this study).
Time Frame: Week 16
Population: Intent-To-Treat Part 1 (ITT Part 1) population comprises all participants who were randomized and received at least one dose of the study medication during Part 1. Results for binary endpoints are based on non-responder imputation (NRI).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: MTX Escalated Dose | Part 1: ADA + MTX
Number analyzed (Participants) | 122 | 123
percentage of participants | 13.1 [7.1 to 19.1] | 41.5 [32.8 to 50.2]
Statistical Analysis 1: Comparison: Part 1: MTX Escalated Dose vs Part 1: ADA + MTX; Test type: Other — Between group difference; p < 0.001, Cochran-Mantel-Haenszel; Adjusted for the stratification factor which is the duration of prior MTX 15 mg ew use of ≤ 3 months or > 3 months; point estimate difference = 28.3, 95% CI 2-sided [17.8 to 38.9]

2. Secondary Outcome: Change in Dermatology Life Quality Index (DLQI) Score From Baseline (Part 1)
Description: The Dermatology Life Quality Index (DLQI) score is a measure of participant's quality of life (QOL) related to skin disease.The DLQI questionnaire consists of 10 questions concerning participants' perception of the impact of skin diseases on different aspects of their health related QOL over the last week. The items of the DLQI encompass aspects such as symptoms and feelings, daily activities, leisure, work or school, personal relationships and the side effects of treatment. The range of possible DLQI scores is 0 to 30, with a score of 0 indicating no effect at all on a participant's life and a score of 30 indicating extremely large effect on participant's life. A decrease in DLQI score indicates improvement.
Time Frame: From Day 1 to Week 16
Population: ITT (Part 1). Results for binary endpoints are based on NRI. Results for other continuous endpoints are based on MMRM.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Part 1: MTX Escalated Dose | Part 1: ADA + MTX
Number analyzed (Participants) | 109 | 117
score on a scale | -3.1 [-3.85 to -2.30] | -5.9 [-6.70 to -5.20]

3. Secondary Outcome: Change in Tender Dactylitic Digit Count From Baseline for Participants With Presence of Dactylitis at Baseline (Part 1)
Description: Hands and feet bilaterally were assessed for the presence/absence of dactylitis and associated tenderness for participants with presence of dactylitis at baseline. The tender dactylitic digit count is equal to the number of swollen and painful digits (range 0 to 20). A decrease indicates improvement.
Time Frame: From Day 1 to Week 16
Population: ITT (Part 1) Results for binary endpoints are based on NRI. Results for other continuous endpoints are based on MMRM.
Measure: Least Squares Mean (95% Confidence Interval); unit: count of fingers/ toes with dactylitis
Arm/Group | Part 1: MTX Escalated Dose | Part 1: ADA + MTX
Number analyzed (Participants) | 66 | 62
count of fingers/ toes with dactylitis | -0.9 [-1.48 to -0.41] | -2.8 [-3.35 to -2.23]

4. Secondary Outcome: Change in Disease Activity Score 28 (DAS28)-C-reactive Protein (CRP) Score From Baseline (Part 1)
Description: The Disease Activity Score 28 (DAS28) is a validated index of rheumatoid arthritis disease activity but is also used in PsA clinical trials. DAS28 is a composite score calculated using a mathematical formula based on the scores for these scales. DAS28 includes tender and swollen joint counts, PtGA, and acute phase reactant (CRP in this study). DAS28 scores range from 0 to 10, with higher scores indicating more disease activity. A larger negative change in the DAS28 score indicates greater improvement.
Time Frame: From Day 1 to Week 16
Population: ITT (Part 1) Results for binary endpoints are based on NRI. Results for other continuous endpoints are based on MMRM.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Part 1: MTX Escalated Dose | Part 1: ADA + MTX
Number analyzed (Participants) | 108 | 114
score on a scale | -0.9 [-1.08 to -0.65] | -2.0 [-2.16 to -1.75]

5. Secondary Outcome: Change in Psoriatic Arthritis Impact of Disease Score (PsAID) Score From Baseline (Part 1)
Description: Psoriatic Arthritis Impact of Disease Score (PsAID) was developed by an European League Against Rheumatism (EULAR) initiative and is a validated patient self-reported tool to assess the impact of PsA on the participant's life. The PsAID is a composite score calculated using a mathematical formula based on the scores for each component. PsAID-9 was developed for clinical trials and was used in this study. The PsAID-9 is calculated based on 9 Numerical rating scales (NRS) questions that include pain, fatigue, skin, work and/or leisure activities, function, discomfort, sleep, coping, and anxiety). Each NRS is assessed as a number between 0 and 10. PsAID scores range from 0 to 10, with higher scores indicating worse status. A larger negative change in the PsAID-9 score indicates greater improvement.
Time Frame: From Day 1 to Week 16
Population: ITT (Part 1) Results for binary endpoints are based on NRI. Results for other continuous endpoints are based on MMRM.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Part 1: MTX Escalated Dose | Part 1: ADA + MTX
Number analyzed (Participants) | 107 | 117
score on a scale | -1.7 [-2.09 to -1.28] | -3.3 [-3.73 to -2.95]

6. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology (ACR) 20/50/70 Response (Part 1)
Description: The ACR is a standard criteria originally developed to measure the effectiveness of various arthritis medications or treatments in clinical trials for RA, but is also widely used in PsA. The ACR measures improvement in tender joint count (TJC) or swollen joint count (SJC), and improvement in at least 3 of the following 5 parameters: Patient Global Assessment (PtGA), Physician's Global Assessment of Disease Activity (PhGA), physical function (using HAQ-DI) and acute phase reactant (using CRP). ACR 20/50/70 response is achieved if ≥ 20%/≥ 50%/≥ 70% improvement in tender joint count (TJC) or swollen joint count (SJC) as well as a ≥ 20%/≥ 50%/≥ 70% improvement in ≥ 3 of the other 5 parameters.
Time Frame: Week 16
Population: ITT (Part 1) Results for binary endpoints are based on NRI. Results for other continuous endpoints are based on MMRM.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: MTX Escalated Dose | Part 1: ADA + MTX
Number analyzed (Participants) | 122 | 123
percentage of participants
  ACR 20 | 32.8 [24.5 to 41.1] | 67.5 [59.2 to 75.8]
  ACR 50 | 16.4 [9.8 to 23.0] | 45.5 [36.7 to 54.3]
  ACR 70 | 8.2 [3.3 to 13.1] | 30.9 [22.7 to 39.1]

7. Secondary Outcome: Change in Leeds Enthesitis Index (LEI) From Baseline (Part 1) for Participants With Presence of LEI at Baseline
Description: The Leeds Enthesitis Index (LEI) is an enthesitis measure developed specifically for PsA and assesses the presence or absence of tenderness at the following 3 bilateral enthesial sites: medial femoral condyles, lateral epicondyles of the humerus, and Achilles tendon insertions for participants with presence of LEI at baseline.Tenderness on examination is recorded as either present (1) or absent (0) for each of the 6 sites, for an overall score range of 0 to 6. A decrease in LEI indicates improvement.
Time Frame: From Day 1 to Week 16
Population: ITT (Part 1) Results for binary endpoints are based on NRI. Results for other continuous endpoints are based on MMRM.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Part 1: MTX Escalated Dose | Part 1: ADA + MTX
Number analyzed (Participants) | 89 | 92
score on a scale | -1.1 [-1.43 to -0.75] | -1.9 [-2.22 to -1.54]

8. Secondary Outcome: Percentage of Participants in MDA in Part 2 of the Study (Week 32)
Description: MDA for PsA was defined as fulfilling at least 5 of the following 7 criteria: TJC ≤ 1 (out of TJC68 assessed in this study), SJC ≤ 1 (out of SJC66 assessed in this study), PASI ≤ 1 or BSA ≤ 3; Patient's assessment of pain VAS ≤ 15, PtGA VAS ≤ 20, HAQ-DI score ≤ 0.5, and tender entheseal points ≤ 1 (out of 8 assessed in this study).
Time Frame: Week 32
Population: ITT Long Term (ITT LT) population comprises all participants who continued to Part 2 and received at least one dose of Part 2 study medication. No missing data imputationperformed for long term efficacy analysis except for participants who were rescued, where participants rescued prior to Week 32 are imputed as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part 2: ADA + MTX Escalated Dose: Participants not achieving MDA at Week 16 on MTX escalated to 20 - 25 mg or highest tolerable dose ew, received adalimumab (ADA) 40 mg every other week (eow) in combination with MTX 20 - 25 mg or highest tolerable dose ew
Arm/Group | Part 2: MTX Escalated Dose | Part 2: ADA + MTX Escalated Dose | Part 2: ADA | Part 2: ADA ew + MTX
Number analyzed (Participants) | 15 | 91 | 51 | 57
percentage of participants | 66.7 [42.8 to 90.5] | 54.9 [44.7 to 65.2] | 80.4 [69.5 to 91.3] | 29.8 [17.9 to 41.7]

9. Secondary Outcome: Change in Psoriatic Arthritis Disease Activity Score (PASDAS) From Baseline (Part 1)
Description: Psoriatic Arthritis Disease Activity Score (PASDAS) is a weighted disease activity measure developed specifically for PsA. It includes PhGA, PtGA, SF-36 PCS, SJC, TJC, Leeds enthesitis count, tender dactylitic count and hsCRP lab test. The PASDAS is a composite score calculated using a mathematical formula based on the scores for each component. The PASDAS is unitless, with a typical score range between 0 and 10. Smaller values on PASDAS indicate a better condition; a negative change from baseline indicates improvement.
  .
Time Frame: From Day 1 to week 16
Population: ITT (Part 1) Results for binary endpoints are based on NRI. Results for other continuous endpoints are based on MMRM.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Part 1: MTX Escalated Dose | Part 1: ADA + MTX
Number analyzed (Participants) | 105 | 114
score on a scale | -1.2 [-1.46 to -0.86] | -2.8 [-3.05 to -2.48]

10. Secondary Outcome: Change in Short Form Health Survey 36 (SF-36) Score From Baseline (Part 1)
Description: The Short Form Health Survey 36 (SF-36) is a generic measure to assess participant's general health/well-being (health related quality of life); short version 2 (SF-36v2) was used. SF-36 determined participants' overall quality of life by assessing 1) limitations in physical functioning due to health problems; 2) limitations in usual role because of physical health problems; 3) bodily pain; 4) general health perceptions; 5) vitality; 6) limitations in social functioning because of physical or emotional problems; 7) limitations in usual role due to emotional problems; and 8) general mental health. Items 1-4 comprise physical component of the SF-36. Scores on each item were summed and averaged (PCS; range = 0-100). Items 5-8 comprise mental component of the SF-36. Scores on each item were summed and averaged (mental component score [MCS]; range = 0-100). Larger values on SF-36 indicate a better condition. A positive change from Baseline in either PCS or MCS indicates improvement.
Time Frame: From Day 1 to Week 16
Population: ITT (Part 1)
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Part 1: MTX Escalated Dose | Part 1: ADA + MTX
Number analyzed (Participants) | 107 | 117
score on a scale
  SF-36 PCS | 4.4 [3.07 to 5.73] | 8.9 [7.58 to 10.15]
  SF-36 MCS | 1.3 [-0.36 to 2.97] | 4.4 [2.85 to 6.05]

11. Secondary Outcome: Change in HAQ-DI Score From Baseline (Part 1)
Description: The HAQ-DI is a standardized measure of physical function in arthritis. The HAQ-DI questionnaire contains 20 items divided into 8 domains that measure: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and common daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where 0 represents no disability and 3 very severe, high-dependency disability. HAQ remission indicating normal physical function is defined by HAQ-DI score of < 0.5. Negative change from Baseline indicates improvement.
Time Frame: From Day 1 to Week 16
Population: ITT (Part 1) Results for binary endpoints are based on NRI. Results for other continuous endpoints are based on MMRM.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Part 1: MTX Escalated Dose | Part 1: ADA + MTX
Number analyzed (Participants) | 110 | 116
score on a scale | -0.3 [-0.39 to -0.21] | -0.5 [-0.60 to -0.42]

12. Secondary Outcome: Percentage of Participants Achieving Psoriasis Area and Severity Index (PASI) 75/90/100 Response Among Participants With BSA Greater Than or Equal to 3% at Baseline (Part 1)
Description: Psoriasis Area and Severity Index (PASI) provides a quantitative assessment of psoriasis lesional burden based on the amount of body surface area involved and the degree of severity of erythema, induration, and scale, weighted by body part. The score ranges from 0 to 72, with 0 indicating no psoriasis and 72 indicating very severe psoriasis. 75/90/100 denotes greater than or equal to 75%/90%/100% improvement in PASI score. A 100% reduction is considered complete clearance of psoriasis.
Time Frame: Week 16
Population: ITT (Part 1) Results for binary endpoints are based on NRI. Results for other continuous endpoints are based on MMRM.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: MTX Escalated Dose | Part 1: ADA + MTX
Number analyzed (Participants) | 87 | 78
percentage of participants
  PASI 75 | 31.0 [21.3 to 40.8] | 73.1 [63.2 to 82.9]
  PASI 90 | 18.4 [10.3 to 26.5] | 57.7 [46.7 to 68.7]
  PASI 100 | 9.2 [3.1 to 15.3] | 29.5 [19.4 to 39.6]

13. Secondary Outcome: Change in Disease Activity in Psoriatic Arthritis Score (DAPSA) Score From Baseline (Part 1)
Description: Disease Activity in Psoriatic Arthritis Score (DAPSA) score is a the sum of swollen joint count (66 joints), tender joint count (68 joints), CRP (mg/dL), Patient's Assessment of Pain (on a 10-unit VAS;0=no pain, 10=worst possible pain), and Patient's Global Assessment of Disease Activity (arthritis, on a 10-unit VAS; 0 to 100 centimeter [cm] VAS, 0=excellent and 10=poor). Change from baseline in DAPSA measures the change in disease activity, where a negative change indicates an improvement and a positive change indicates worsening of disease activity.
Time Frame: From Day 1 to Week 16
Population: ITT (Part 1) Results for binary endpoints are based on NRI. Results for other continuous endpoints are based on MMRM.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Part 1: MTX Escalated Dose | Part 1: ADA + MTX
Number analyzed (Participants) | 108 | 114
score on a scale | -12.1 [-15.57 to -8.69] | -28.2 [-31.60 to -24.87]

ADVERSE EVENTS:
Time Frame: All adverse events reported from the time of study medication administration until 70 days following discontinuation of study medication administration have elapsed.
Description: The Safety population Part 1 included all participants who received at least 1 dose of Part 1 study medication (1 of the 2 treatment arms) and in Part 2, all participants who received at least 1 dose of Part 2 study medication (1 of 4 treatment arms).
  Two sets of safety analyses performed using the Safety Population Part 1 and Safety Population Part 2, respectively:
  * Safety analyses during Part 1 (up to Week 16).
  * Safety analyses during Part 2 (Week 16 to Week 32).
Groups:
- Part 1: MTX Escalated Dose: Methotrexate (MTX) escalated to 20 - 25 mg or highest tolerable dose every week (ew) (MTX 20 - 25 mg or highest tolerable dose ew)
- Part 1: ADA + MTX: Adalimumab (ADA) 40 mg every other week (eow) in combination with MTX 15 mg ew (ADA 40 mg eow + MTX 15 mg ew
- Part 2: MTX Escalated Dose: Participants achieving MDA at Week 16 on MTX escalated to 20 -25 mg or highest tolerable dose ew, continued with the same MTX dose (MTX 20 - 25 mg or highest tolerable dose ew)
- Part 2: ADA + MTX Escalated Dose: Participants not achieving MDA at Week 16 on MTX escalated to 20 - 25 mg or highest tolerable dose ew, received ADA 40 mg eow in combination with MTX 20 - 25 mg or highest tolerable dose ew (ADA 40 mg eow plus MTX 20 - 25 mg or highest tolerable dose ew)
- Part 2: ADA: Participants achieving MDA at Week 16 on ADA 40 mg eow plus MTX 15 mg ew, had MTX completely withdrawn at Week 16 and continued receiving ADA as monotherapy (ADA 40 mg eow),
- Part 2: ADA ew + MTX: Participants not achieving MDA at Week 16 on ADA 40 mg eow plus MTX 15 mg ew, had ADA escalated to 40 mg ew in combination with MTX 15 mg ew (ADA 40 mg ew plus MTX 15 mg ew)
Arm/Group | Part 1: MTX Escalated Dose | Part 1: ADA + MTX | Part 2: MTX Escalated Dose | Part 2: ADA + MTX Escalated Dose | Part 2: ADA | Part 2: ADA ew + MTX
All-Cause Mortality (participants affected / at risk) | 0/122 | 0/123 | 0/15 | 0/95 | 0/54 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/122 | 2/123 | 0/15 | 3/95 | 1/54 | 3/63
Other Adverse Events (participants affected / at risk) | 32/122 | 24/123 | 5/15 | 25/95 | 5/54 | 20/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: MTX Escalated Dose (N=122) | Part 1: ADA + MTX (N=123) | Part 2: MTX Escalated Dose (N=15) | Part 2: ADA + MTX Escalated Dose (N=95) | Part 2: ADA (N=54) | Part 2: ADA ew + MTX (N=63)
GASTRIC MUCOSA ERYTHEMA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SCIATICA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URETEROLITHIASIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UTERINE POLYP (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: MTX Escalated Dose (N=122) | Part 1: ADA + MTX (N=123) | Part 2: MTX Escalated Dose (N=15) | Part 2: ADA + MTX Escalated Dose (N=95) | Part 2: ADA (N=54) | Part 2: ADA ew + MTX (N=63)
NAUSEA (Gastrointestinal disorders) | 11 (13) | 5 (5) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
DRUG INTOLERANCE (General disorders) | 8 (12) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEPATITIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 1 (1) | 2 (2)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 11 (11) | 10 (10) | 0 (0) | 13 (13) | 2 (2) | 9 (11)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 1 (2) | 3 (5)
TRANSAMINASES INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4)
PSORIATIC ARTHROPATHY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 4 (4)
HEADACHE (Nervous system disorders) | 2 (3) | 10 (10) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 7 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2019-06-03): https://cdn.clinicaltrials.gov/large-docs/75/NCT02814175/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-10): https://cdn.clinicaltrials.gov/large-docs/75/NCT02814175/SAP_001.pdf